CLINICAL TRIAL: NCT01165632
Title: A Pilot Study of Utility of 18F-FDOPA-PET for Neurosurgical Planning and Radiotherapy Target Delineation in Glioma Patients: Biopsy Validation of 18F-FDOPA-PET Uptake and Biodistribution in Brain Tumors
Brief Title: Fluorine F 18 Fluorodopa-Labeled PET Scan in Planning Surgery and Radiation Therapy in Treating Patients With Newly Diagnosed High- or Low-Grade Malignant Glioma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MC1078; NCI-2010-01607 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-001904 (Other: Mayo Clinic IRB); MC1078 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2010-07-14; First posted 2010-07-20 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Diffuse Astrocytoma; Adult Ependymoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Adult Myxopapillary Ependymoma; Adult Oligodendroglioma; Adult Pilocytic Astrocytoma; Adult Pineal Gland Astrocytoma; Adult Subependymal Giant Cell Astrocytoma; Adult Subependymoma
MeSH Terms: conditions — Astrocytoma; Ependymoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Glioma, Subependymal | interventions — Biopsy; Radiotherapy; Radiation; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; fluorodopa F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Beginning at no more than 1 week before biopsy or resection, patients undergo fluorine F 18 fluorodopa-labeled PET/CT scan and pre-operative MRI. Patients then undergo stereotactic craniotomy. Some patients may also undergo radiation therapy.
  Interventions: Procedure: biopsy; Procedure: computed tomography; Procedure: therapeutic conventional surgery; Radiation: radiation therapy treatment planning/simulation; Radiation: radiation therapy; Procedure: magnetic resonance imaging; Procedure: positron emission tomography; Drug: fluorine F 18 fluorodopa

INTERVENTIONS:
Procedure: biopsy — Correlative studies
  Other Names: biopsies
Procedure: computed tomography — Undergo computed tomography
  Other Names: tomography, computed
Procedure: therapeutic conventional surgery — Undergo stereotactic craniotomy
Radiation: radiation therapy treatment planning/simulation — Undergo radiation therapy treatment planning/simulation
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Procedure: magnetic resonance imaging — Undergo magnetic resonance imaging
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Procedure: positron emission tomography — Undergo positron emission tomography
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Drug: fluorine F 18 fluorodopa — Given IV
  Other Names: (18)F-FDOPA; 18F-6- L-fluorodopa; 18F-DOPA; 18F-FDOPA

SUMMARY:
RATIONALE: New imaging procedures, such as fluorine F 18 fluorodopa-labeled PET scan, may help in guiding surgery and radiation therapy and allow doctors to plan better treatment.

PURPOSE: This clinical trial studies fluorine F 18 fluorodopa-labeled PET scan in planning surgery and radiation therapy in treating patients with newly diagnosed high- or low-grade malignant glioma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine correlation between 18F-FDOPA PET activity, MRI contrast enhancement, and high- or low-grade glioma biopsies.

II. To compare radiotherapy target volume delineation with and without 18F- FDOPA-PET metabolic imaging information to determine role of metabolic imaging in radiotherapy treatment planning.

SECONDARY OBJECTIVES:

I. To determine correlation between concordance of 18F-FDOPA PET activity, MRI contrast enhancement, and high- or low-grade glioma biopsies and patient outcomes including overall survival and progression free survival.

OUTLINE:

Beginning at no more than 1 week before biopsy and resection, patients undergo fluorine F 18 fluorodopa-labeled PET/CT scan and pre-operative MRI. Patients then undergo stereotactic craniotomy. Some patients may also undergo radiation therapy.

After completion of study treatment, patients are followed up every year for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* MRI findings compatible with newly diagnosed high- or low-grade malignant glioma
* Planned craniotomy and resection or biopsy
* Willing to sign release of information for any radiation and/or follow-up records
* Negative pregnancy test done =< 48 hours of injection of study drug, for women of childbearing potential only
* Provide informed written consent
* Patients with eGFR < 60 mg/min/1.72m2 are eligible for the study; PLEASE NOTE: the patient is not eligible to receive the contrast for the pMRI at the study dose.

Exclusion Criteria:

* Unable to undergo MRI scans with contrast (e.g. cardiac pacemaker, defibrillator, kidney failure)
* Unable to undergo an 18F-FDOPA PET scan (e.g. Parkinson's Disease, taking anti-dopaminergic, or dopamine agonist medication or less than 6 half-lives from discontinuance of dopamine agonists)
* Pregnant women; nursing women; men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07-26 (Actual); Primary Completion 2013-11-05 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
18F-FDOPA PET activity, MRI contrast enhancement, and high- or low-grade glioma biopsies | Up to 2 years
  Determine correlation between 18F-FDOPA PET activity, MRI contrast enhancement, and high- or low-grade glioma biopsies.
18F- FDOPA-PET metabolic imaging information | Up to 2 years
  Compare radiotherapy target volume delineation with and without 18F- FDOPA-PET metabolic imaging information to determine role of metabolic imaging in radiotherapy treatment planning.

SECONDARY OUTCOMES:
Concordance of 18F-FDOPA PET and 11C-choline activity, MRI contrast enhancement, and high- or low-grade glioma biopsies | Up to 2 years
  Determine correlation between concordance of 18F-FDOPA PET and 11C-choline activity, MRI contrast enhancement, and high- or low-grade glioma biopsies and patient outcomes including overall survival and progression free survival.
With and without 18F- FDOPA PET, 11C-choline PET metabolic imaging information | 2 Years
  Compare radiotherapy target volume delineation with and without 18F- FDOPA PET, 11C-choline PET metabolic imaging information; pMRI and DTI advanced MR imaging, to determine role in radiotherapy treatment planning.
18F-FDOPA PET activity, 11C-choline PET activity, MRI contrast enhancement, pMRI, and DTI, with high- or low-grade glioma biopsies | 2 years
  Determine correlation between 18F-FDOPA PET activity, 11C-choline PET activity, MRI contrast enhancement, pMRI, and DTI, with high- or low-grade glioma biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N. Laack, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials